CLINICAL TRIAL: NCT01805882
Title: A Pilot Study to Evaluate the Safety and Efficacy of Multiple Anti-HCV Combination Therapy in Chronically Infected Hepatitis C Patients
Brief Title: Combination Therapy for Chronic Hepatitis C Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130066; 13-I-0066 (Other: NIH)
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis C, Chronic
Keywords: Interferon Sparing; Directly Acting Antiviral; Ribavarin Sparing
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir; ledipasvir; GS-9669; GS-9451

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- A: HCV GT-1, tx naïve, 12 wks Sofosbuvir/Ledipasvir (Experimental): Oral treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885), once daily, for 12 weeks in HCV genotype 1, treatment naïve patients
  Interventions: Drug: Sofosbuvir; Drug: Ledipasvir
- B: HCV GT-1, tx naïve, 6 wks Sofosbuvir/Ledipasvir/GS-9669 (Experimental): Oral treatment with Sofosbuvir 400mg (GS-7977), Ledipasvir 90mg (GS-5885), GS-9669 500mg, once daily, for 6 weeks in HCV genotype 1, treatment naïve patients
  Interventions: Drug: Sofosbuvir; Drug: Ledipasvir; Drug: GS-9669
- C: HCV GT-1, tx naïve, 6 wks Sofosbuvir/Ledipasvir/GS-9451 (Experimental): Oral treatment with Sofosbuvir 400mg (GS-7977), Ledipasvir 90mg (GS-5885), GS-9451 80mg, once daily, for 6 weeks in HCV genotype 1, treatment naïve patients
  Interventions: Drug: Sofosbuvir; Drug: Ledipasvir; Drug: GS-9451
- D: HCV GT-1, tx-relapsed, 12 wks Sofosbuvir/Ledipasvir (Experimental): Oral treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885), once daily, for 12 weeks in HCV genotype 1, treatment-relapsed patients who previously received Sofosbuvir plus Ribavirin
  Interventions: Drug: Sofosbuvir; Drug: Ledipasvir
- E: HCV GT-4, tx naïve/expd, 12 wks Sofosbuvir/Ledipasvir (Experimental): Oral treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885), once daily, 12 weeks in HCV genotype 4 treatment naïve subjects and interferon treament experienced subjects
  Interventions: Drug: Sofosbuvir; Drug: Ledipasvir
- F: HCV GT-1, tx naïve/expd 6 wks Sofosbuvir/Ledipasvir/GS-9451 (Experimental): Oral treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885) and GS-9451 80mg, once daily, 6 weeks in HCV genotype 1 treatment naïve and treatment experienced subjects with advanced liver disease
  Interventions: Drug: Sofosbuvir; Drug: Ledipasvir; Drug: GS-9451
- G: HCV GT-1, tx naïve, 4 wks Sofosbuvir, Ledipasvir, GS-9451 (Experimental): Oral Treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885) with GS-9451 80mg, once daily, 4 weeks in HCV genotype 1 treatment naïve subjects with early stage liver disease
  Interventions: Drug: Sofosbuvir; Drug: Ledipasvir; Drug: GS-9451
- H: HCV GT-1, tx naïve, 4 wks Sofos/Ledip/GS-9451/GS-9669 (Experimental): Oral Treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885) with GS-9451 80mg, and GS-9669 250mg, once daily, 4 weeks in HCV genotype 1 treatment naïve subjects with early stage liver disease
  Interventions: Drug: Sofosbuvir; Drug: Ledipasvir; Drug: GS-9669; Drug: GS-9451
- D Retx: HCV GT-1, Re-Treatment, 12 wks Sofosbuvir, Ledipasvir (Experimental): Oral treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885), once daily, 12 weeks in HCV genotype 1 subjects who failed HCV therapy in Arm B or Arm G or Arm H
  Interventions: Drug: Sofosbuvir; Drug: Ledipasvir

INTERVENTIONS:
Drug: Sofosbuvir
  Other Names: Sofosbuvir (GS-7977)
Drug: Ledipasvir
  Other Names: Ledipasvir (GS-5885)
Drug: GS-9669
  Arms: B: HCV GT-1, tx naïve, 6 wks Sofosbuvir/Ledipasvir/GS-9669; H: HCV GT-1, tx naïve, 4 wks Sofos/Ledip/GS-9451/GS-9669
Drug: GS-9451
  Arms: C: HCV GT-1, tx naïve, 6 wks Sofosbuvir/Ledipasvir/GS-9451; F: HCV GT-1, tx naïve/expd 6 wks Sofosbuvir/Ledipasvir/GS-9451; G: HCV GT-1, tx naïve, 4 wks Sofosbuvir, Ledipasvir, GS-9451; H: HCV GT-1, tx naïve, 4 wks Sofos/Ledip/GS-9451/GS-9669

SUMMARY:
Background:

- GS-7977, GS-5885, GS-9669, and GS-9451 are new drugs for treating hepatitis C virus (HCV) infection. GS-7977 may help treat the infection when used with other treatments like interferon therapy. GS-5885, and GS-9669, and GS-9451 also lower the amount of HCV in the body. Researchers want to see whether GS-7977 can be combined with any of the other three drugs to treat HCV infection. Some participants will take GS-7977 and GS-5885. Others will take GS-7977, GS-5885 and GS-9669 or GS-7977, GS-5885 and GS-9451.

Objectives:

- To see whether GS-7977 with GS-5885 alone or in combination with either GS-9669 or 9451 can be used to treat HCV infection.

Eligibility:

Individuals at least 18 years of age who have chronic HCV infection and have never been treated for it.

Individuals at least 18 years of age who have chronic HCV infection and have not responded to interferon therapy.

Individuals at least 18 years of age who have chronic HCV infection with advanced liver disease and have never been treated for HCV

Design:

Participants will be screened with a physical exam and medical history. Blood samples will be collected. A liver biopsy may also be performed.

Some participants will take the two study drugs and some will take three study drugs. Those who take GS-7977 and GS-5885 will have one daily tablet named fixed dose combination or FDC. Those who take GS-7977 and CS-9669 will have three daily tablets taken once daily. Those who take GS-7977 and GS-5885 and GS-9451 will take 2 pills once a day. GS-7977 and GS-5885 will be combined in one pill and GS-9451 will be in another pill.

Treatment will be monitored with frequent blood tests. These tests will check liver function and the level of HCV infection. Participants may have other blood tests as needed for treatment.

Participants will have 4, 6 or 12 weeks of treatment depending on which study drugs are scheduled to take. After they complete their schedule, they will stop treatment with the study drugs. They may also have another liver biopsy.

Participants will have regular follow-up visits over the next 48 weeks. They will have physical exams and provide blood samples....

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is a major public health problem with an estimated 180 million people infected worldwide. In the United States an estimated 4.1 million people are infected, and HCV is the principal cause of death from liver disease and leading indication for liver transplantation. While treatment with ribavirin (RBV) and pegylated interferon (PEG) in combination with boceprevir/telaprevir is the currently recommended therapy for chronic HCV infection and has superior cure rates compared to PEG+RBV alone in HCV monoinfected patients, treatment is still associated with a high incidence of adverse events (AEs), discontinuations, and poor cure rates in several populations. Recent studies have demonstrated that the use of a combination of antivirals, which target HCV without interferon (IFN), can cure HCV without additional toxicities. However, the determinants of response to IFN-free regimens have not been established.

This is an open label study to assess the safety, tolerability, and efficacy of treatment with GS-7977 with GS-5885, alone or in combination with GS-9669 and/or GS-9451 (selective HCV nucleotide NS5B, NS5A, nonnucleotide NS5B and NS3 inhibitors, respectively) in HCV infected treatment naive and treatment experienced patients with early and advanced liver disease. The findings from this study will aid in our understanding of determinants of response to an IFN-free regimen in HCV infected patients for both patients with early and advanced liver disease as well as in patients who are treatment naive and those who have been treated before for HCV.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Eighteen years of age or older at screening.
  2. Female study participants with childbearing potential (as defined below) and all males must be willing to practice either:

     * Abstinence from sexual intercourse or
     * One or more forms of effective barrier contraception throughout dosing and for 30 days following the last dose. This cannot include hormonal contraception for female subjects.

     Effective forms of barrier contraception include:
     * a male condom with spermicide
     * use by female sexual partner of a female condom with spermicide

     Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) includes any female who:
     * Has had a hysterectomy or
     * Has had a bilateral oophorectomy (ovariectomy) or
     * Is post-menopausal (a demonstration of a total cessation of menses for greater than or equal to1 year)
     * Has had a bilateral tubal ligation or fallopian tube inserts
  3. Chronic HCV GT-1 or GT-4 infection as documented by greater than or equal to 1 measurement of serum HCV RNA greater than or equal to 2,000 international units per milliliter during screening and at least one of the following:

     * A positive anti-HCV antibody, HCV RNA, or HCV genotype test result greater than or equal to 12 months prior to the baseline (day 0) visit together with current positive HCV RNA and anti-HCV antibody test results or
     * Positive HCV RNA test and anti-HCV antibody test results together with a liver biopsy consistent with chronic HCV infection or a liver biopsy performed before enrollment with evidence of chronic hepatitis C infection disease, such as the presence of fibrosis.
  4. Group A may include up to 20% of subjects with compensated cirrhosis.

     Group B and C may only include subjects with absence of cirrhosis.

     Group D, D-ReTx & E may include subjects with compensated cirrhosis.

     Group F may only include patients with advanced liver disease (historic Metavir or HAI Stage 3 or 4 or ISHAK Stage 4, 5 or 6 or cirrhosis as defined below)

     Group G and H may only include those with absence of cirrhosis and HAI Stage 0-2 or FibroTest as below.

     Cirrhosis is defined as any one of the following:
     1. Any biopsy showing cirrhosis.
     2. A FibroTest(r) score of greater than or equal to 0.75 AND an AST: platelet ratio (APRI) of > 2 performed within 12 months of screening.

     Liver imaging within 6 months of Day 0 to exclude hepatocellular carcinoma (HCC) is required in patients with cirrhosis.

     Absence of cirrhosis is defined as one of the following:
     1. A liver biopsy performed within 36 calendar months of screening showing absence of cirrhosis.
     2. A FibroTest(r) score of < 0.48 AND APRI of < 1 performed within 6 months of screening. This would also qualify a subject for Group G and H as having Stage 0-2 disease in the absence of a liver biopsy.

     In the absence of a definitive diagnosis of presence or absence of cirrhosis by the above criteria, a liver biopsy is required (for Groups B, C, G and H).
  5. Ability to communicate effectively with the study investigator and other key personnel.
  6. Willing to give written informed consent and comply with the study restrictions and requirements.
  7. Opioid-dependent individuals must be participating in a supervised treatment program.
  8. Subjects must have an external primary care doctor (outside of the CC and the NIH) for their medical management.

EXCLUSION CRITERIA:

1. Current or prior history of any of the following:

   * Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol; subjects currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded.
   * Gastrointestinal disorder or post operative condition that could interfere with the absorption of the study drug.
   * Poor venous access interfering with required study blood collection.
   * Clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage).
   * Solid organ transplantation.
   * Significant pulmonary disease, significant cardiac disease or porphyria.
   * Unstable psychiatric disease (Subjects with psychiatric illness that is well-controlled on a stable treatment regimen or currently not requiring medication may be included).
   * Any malignancy or its treatment that in the opinion of the PI may cause ongoing interference with host immunity; subjects under evaluation for malignancy are not eligible.
   * Significant drug allergy (such as anaphylaxis or hepatotoxicity).
   * Substance abuse, which in the opinion of the investigator is likely to interfere with medication adherence or study compliance.
   * Lactose allergy, patients with lactose intolerance will be evaluated on a case-by-case basis.
2. Positive test results at screening for hepatitis B virus (HBV) surface antigen (HBsAg), HBV DNA (if medically indicated) or anti-HIV antibody (unless previously treated on 13-I-0159).
3. Prior exposure to any direct-acting antivirals for HCV infection, except for patients who were previously treated studies 11-I-0258, 13-I-1059 or this study enrolling in Group D.
4. History of clinically significant chronic liver disease due to other etiology (e.g., hemochromatosis, autoimmune hepatitis, Wilson s disease, alpha 1-antitrypsin deficiency, alcoholic liver disease, > moderate non-alcoholic steatohepatitis and toxin exposures).
5. Use of herbal/natural remedies for potential benefit to the liver within 21 Days of Day 0.
6. History of ascites, variceal hemorrhage, hepatic encephalopathy, or conditions consistent with decompensated liver disease.
7. Screening or baseline ECG with clinically significant ECG findings, or a personal/first degree relative history of Torsade de pointes.
8. Abnormal hematological and biochemical parameters at screening, including:

   * Neutrophil count less than 750 cells per cubic millimeter.
   * Hemoglobin level < 9 g/dL. If Hgb < 11g/dL in women and < 12 g/dL in men other causes of anemia should be excluded as medically indicated.
   * Platelet count less than or equal to 50,000 cells per cubic millimeter.
   * Estimated glomerular filtration rate less than 50 milliliter/min/1.73m(2).
   * ALT or AST level greater than or equal to 10 times upper limit of normal (ULN).
   * Serum lipase level greater than or equal to 1.5 times upper limit of normal (ULN)at screening or during the screening period in a patient with symptoms consistent with pancreatitis.
   * Total bilirubin level greater than or equal to 2.0 times upper limit of normal (ULN), except in subjects with Gilbert s syndrome.
   * Albumin level less than or equal to 3.0 grams per deciliter in patients without cirrhosis, albumin less than or equal to 2.8 g/dL in cirrhotic patients.
9. Poorly controlled diabetes mellitus indicated by hemoglobin A1C greater than 9% at screening.
10. Donation or loss of blood of greater than 400 milliliter within 8 weeks prior to the first dose of the study drugs.
11. Known hypersensitivity to GS-5885, GS-7977, GS-9669, GS-9451 or formulation excipients.
12. Pregnant/Breastfeeding women.
13. Need for use of the following medications from 21 days prior to the start of study drugs through the end of treatment (unless otherwise specified):

    * Hematologic stimulating agents (e.g. erythropoiesis-stimulating agents (ESAs); granulocyte colony stimulating factor (GCSF); thrombopoietin (TPO) mimetics).
    * Chronic systemic immunosuppressants including, but not limited to, corticosteroids (prednisone equivalent of greater than 10 milligrams per day for greater than 2 weeks), azathioprine, or monoclonal antibodies (e.g., infliximab).
    * Investigational agents or devices for any indication.
    * Medications for disease conditions excluded from the protocol (e.g., active cancer, transplantation) are not listed under this Concomitant Medication section and are disallowed in the study.
    * Concomitant use of certain medications or herbal/natural supplements per PI discretion expected to result in pharmacokinetic interactions resulting in increases or decreases in exposure of study drug(s).
14. Co-enrollment Guidelines: Co-enrollment in other clinical trials is restricted, other than enrollment in observational studies. Study staff should be notified of co-enrollment status, as it may require prior approval of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Masur, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (3):
- United States (3):
  - Unity Health Care, Inc./DC General, Washington D.C., District of Columbia
  - Family Medical and Conseling Services, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
The NIH Biomedical Translational Research Information System

REFERENCES:
- [Background] Armstrong GL, Wasley A, Simard EP, McQuillan GM, Kuhnert WL, Alter MJ. The prevalence of hepatitis C virus infection in the United States, 1999 through 2002. Ann Intern Med. 2006 May 16;144(10):705-14. doi: 10.7326/0003-4819-144-10-200605160-00004. PMID 16702586
- [Background] Serfaty L, Aumaitre H, Chazouilleres O, Bonnand AM, Rosmorduc O, Poupon RE, Poupon R. Determinants of outcome of compensated hepatitis C virus-related cirrhosis. Hepatology. 1998 May;27(5):1435-40. doi: 10.1002/hep.510270535. PMID 9581703
- [Background] Davis GL, Albright JE, Cook SF, Rosenberg DM. Projecting future complications of chronic hepatitis C in the United States. Liver Transpl. 2003 Apr;9(4):331-8. doi: 10.1053/jlts.2003.50073. PMID 12682882
- [Derived] Townsend K, Petersen T, Gordon LA, Kohli A, Nelson A, Seamon C, Gross C, Tang L, Osinusi A, Polis MA, Masur H, Kottilil S. Effect of HIV co-infection on adherence to a 12-week regimen of hepatitis C virus therapy with ledipasvir and sofosbuvir. AIDS. 2016 Jan;30(2):261-6. doi: 10.1097/QAD.0000000000000903. PMID 26691547
- [Derived] Petersen T, Townsend K, Gordon LA, Sidharthan S, Silk R, Nelson A, Gross C, Calderon M, Proschan M, Osinusi A, Polis MA, Masur H, Kottilil S, Kohli A. High adherence to all-oral directly acting antiviral HCV therapy among an inner-city patient population in a phase 2a study. Hepatol Int. 2016 Mar;10(2):310-9. doi: 10.1007/s12072-015-9680-7. Epub 2015 Nov 26. PMID 26612014
- [Derived] Kohli A, Kattakuzhy S, Sidharthan S, Nelson A, McLaughlin M, Seamon C, Wilson E, Meissner EG, Sims Z, Silk R, Gross C, Akoth E, Tang L, Price A, Jolley TA, Emmanuel B, Proschan M, Teferi G, Chavez J, Abbott S, Osinusi A, Mo H, Polis MA, Masur H, Kottilil S. Four-Week Direct-Acting Antiviral Regimens in Noncirrhotic Patients With Hepatitis C Virus Genotype 1 Infection: An Open-Label, Nonrandomized Trial. Ann Intern Med. 2015 Dec 15;163(12):899-907. doi: 10.7326/M15-0642. Epub 2015 Nov 24. PMID 26595450
- [Derived] Wilson EM, Kattakuzhy S, Sidharthan S, Sims Z, Tang L, McLaughlin M, Price A, Nelson A, Silk R, Gross C, Akoth E, Mo H, Subramanian GM, Pang PS, McHutchison JG, Osinusi A, Masur H, Kohli A, Kottilil S. Successful Retreatment of Chronic HCV Genotype-1 Infection With Ledipasvir and Sofosbuvir After Initial Short Course Therapy With Direct-Acting Antiviral Regimens. Clin Infect Dis. 2016 Feb 1;62(3):280-288. doi: 10.1093/cid/civ874. Epub 2015 Oct 31. PMID 26521268
- [Derived] Kohli A, Kapoor R, Sims Z, Nelson A, Sidharthan S, Lam B, Silk R, Kotb C, Gross C, Teferi G, Sugarman K, Pang PS, Osinusi A, Polis MA, Rustgi V, Masur H, Kottilil S. Ledipasvir and sofosbuvir for hepatitis C genotype 4: a proof-of-concept, single-centre, open-label phase 2a cohort study. Lancet Infect Dis. 2015 Sep;15(9):1049-1054. doi: 10.1016/S1473-3099(15)00157-7. Epub 2015 Jul 14. PMID 26187031
- [Derived] Kohli A, Osinusi A, Sims Z, Nelson A, Meissner EG, Barrett LL, Bon D, Marti MM, Silk R, Kotb C, Gross C, Jolley TA, Sidharthan S, Petersen T, Townsend K, Egerson D, Kapoor R, Spurlin E, Sneller M, Proschan M, Herrmann E, Kwan R, Teferi G, Talwani R, Diaz G, Kleiner DE, Wood BJ, Chavez J, Abbott S, Symonds WT, Subramanian GM, Pang PS, McHutchison J, Polis MA, Fauci AS, Masur H, Kottilil S. Virological response after 6 week triple-drug regimens for hepatitis C: a proof-of-concept phase 2A cohort study. Lancet. 2015 Mar 21;385(9973):1107-13. doi: 10.1016/S0140-6736(14)61228-9. Epub 2015 Jan 13. PMID 25591505
- [Derived] Osinusi A, Kohli A, Marti MM, Nelson A, Zhang X, Meissner EG, Silk R, Townsend K, Pang PS, Subramanian GM, McHutchison JG, Fauci AS, Masur H, Kottilil S. Re-treatment of chronic hepatitis C virus genotype 1 infection after relapse: an open-label pilot study. Ann Intern Med. 2014 Nov 4;161(9):634-8. doi: 10.7326/M14-1211. PMID 25364884

RESULTS

PARTICIPANT FLOW:
Groups:
- A: HCV GT-1, tx Naive, 12 Wks Sofosbuvir/Ledipasvir: Oral treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885), once daily, for 12 weeks in HCV genotype 1, treatment naïve patients
- B: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9669: Oral treatment with Sofosbuvir 400mg (GS-7977), Ledipasvir 90mg (GS-5885), GS-9669 500mg, once daily, for 6 weeks in HCV genotype 1, treatment naïve patients
- C: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9451: Oral treatment with Sofosbuvir 400mg (GS-7977), Ledipasvir 90mg (GS-5885), GS-9451 80mg, once daily, for 6 weeks in HCV genotype 1, treatment naïve patients
- E: HCV GT-4, tx Naive/Expd, 12 Wks Sofosbuvir/Ledipasvir: Oral treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885), once daily, 12 weeks in HCV genotype 4 treatment naïve subjects and interferon treament experienced subjects
- F: HCV GT-1, tx Naive/Expd 6 Wks Sofosbuvir/Ledipasvir/GS-9451: Oral treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885) and GS-9451 80mg, once daily, 6 weeks in HCV genotype 1 treatment naïve and treatment experienced subjects with advanced liver disease
- G: HCV GT-1, tx Naive, 4 Wks Sofosbuvir, Ledipasvir, GS-9451: Oral Treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885) with GS-9451 80mg, once daily, 4 weeks in HCV genotype 1 treatment naïve subjects with early stage liver disease
- H: HCV GT-1, tx Naive, 4 Wks Sofos/Ledip/GS-9451/GS-9669: Oral Treatment with Sofosbuvir 400mg (GS-7977) and Ledipasvir 90mg (GS-5885) with GS-9451 80mg, and GS-9669 250mg, once daily, 4 weeks in HCV genotype 1 treatment naïve subjects with early stage liver disease
Period: Overall Study
Arm/Group | A: HCV GT-1, tx Naive, 12 Wks Sofosbuvir/Ledipasvir | B: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9669 | C: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9451 | D Retx: HCV GT-1, Re-Treatment, 12 Wks Sofosbuvir, Ledipasvir | D: HCV GT-1, Tx-relapsed, 12 Wks Sofosbuvir/Ledipasvir | E: HCV GT-4, tx Naive/Expd, 12 Wks Sofosbuvir/Ledipasvir | F: HCV GT-1, tx Naive/Expd 6 Wks Sofosbuvir/Ledipasvir/GS-9451 | G: HCV GT-1, tx Naive, 4 Wks Sofosbuvir, Ledipasvir, GS-9451 | H: HCV GT-1, tx Naive, 4 Wks Sofos/Ledip/GS-9451/GS-9669
Started | 20 | 20 | 20 | 34 | 14 | 21 | 50 | 25 | 25
Completed | 20 | 20 | 19 | 32 | 14 | 20 | 48 | 25 | 24
Not Completed | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: HCV GT-1, tx Naive, 12 Wks Sofosbuvir/Ledipasvir | B: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9669 | C: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9451 | D Retx: HCV GT-1, Re-Treatment, 12 Wks Sofosbuvir, Ledipasvir | D: HCV GT-1, Tx-relapsed, 12 Wks Sofosbuvir/Ledipasvir | E: HCV GT-4, tx Naive/Expd, 12 Wks Sofosbuvir/Ledipasvir | F: HCV GT-1, tx Naive/Expd 6 Wks Sofosbuvir/Ledipasvir/GS-9451 | G: HCV GT-1, tx Naive, 4 Wks Sofosbuvir, Ledipasvir, GS-9451 | H: HCV GT-1, tx Naive, 4 Wks Sofos/Ledip/GS-9451/GS-9669 | Total
Number analyzed (Participants) | 20 | 20 | 20 | 34 | 14 | 21 | 50 | 25 | 25 | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 19 | 27 | 11 | 19 | 48 | 24 | 19 | 205
  >=65 years | 1 | 1 | 1 | 7 | 3 | 2 | 2 | 1 | 6 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 4 | 6 | 1 | 7 | 17 | 8 | 6 | 63
  Male | 14 | 12 | 16 | 28 | 13 | 14 | 33 | 17 | 19 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 5
  Not Hispanic or Latino | 19 | 20 | 20 | 34 | 14 | 21 | 46 | 24 | 25 | 223
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 19 | 18 | 28 | 13 | 9 | 29 | 19 | 19 | 169
  White | 3 | 1 | 2 | 5 | 1 | 11 | 17 | 4 | 5 | 49
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Achieve Sustained Viral Response (SVR12) 12 Weeks After the Stop of Treatment Drugs
Description: The primary outcome was the proportion of patients with sustained viral response measured 12 weeks after the stop of treatment. The viral response was assessed by serum HCV RNA concentrations lower than 43 IU/mL - the lower limit of quantification.
Time Frame: 12 weeks after stop of treatment
Population: Subjects who received treatment drugs per arm as listed in the Outcome Measure Description
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | A: HCV GT-1, tx Naive, 12 Wks Sofosbuvir/Ledipasvir | B: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9669 | C: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9451 | D Retx: HCV GT-1, Re-Treatment, 12 Wks Sofosbuvir, Ledipasvir | D: HCV GT-1, Tx-relapsed, 12 Wks Sofosbuvir/Ledipasvir | E: HCV GT-4, tx Naive/Expd, 12 Wks Sofosbuvir/Ledipasvir | F: HCV GT-1, tx Naive/Expd 6 Wks Sofosbuvir/Ledipasvir/GS-9451 | G: HCV GT-1, tx Naive, 4 Wks Sofosbuvir, Ledipasvir, GS-9451 | H: HCV GT-1, tx Naive, 4 Wks Sofos/Ledip/GS-9451/GS-9669
Number analyzed (Participants) | 20 | 20 | 20 | 34 | 14 | 21 | 50 | 25 | 25
percentage of subjects | 100 [83 to 100] | 95 [75 to 100] | 95 [75 to 100] | 91.2 [76 to 98] | 100 [83 to 100] | 95 [76 to 100] | 76 [60 to 85] | 40 [21 to 61] | 20 [7 to 41]

ADVERSE EVENTS:
Arm/Group | A: HCV GT-1, tx Naive, 12 Wks Sofosbuvir/Ledipasvir | B: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9669 | C: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9451 | D Retx: HCV GT-1, Re-Treatment, 12 Wks Sofosbuvir, Ledipasvir | D: HCV GT-1, Tx-relapsed, 12 Wks Sofosbuvir/Ledipasvir | E: HCV GT-4, tx Naive/Expd, 12 Wks Sofosbuvir/Ledipasvir | F: HCV GT-1, tx Naive/Expd 6 Wks Sofosbuvir/Ledipasvir/GS-9451 | G: HCV GT-1, tx Naive, 4 Wks Sofosbuvir, Ledipasvir, GS-9451 | H: HCV GT-1, tx Naive, 4 Wks Sofos/Ledip/GS-9451/GS-9669
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 2/20 | 1/34 | 1/14 | 0/21 | 2/50 | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 17/20 | 20/20 | 20/20 | 34/34 | 14/14 | 17/21 | 48/50 | 24/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: HCV GT-1, tx Naive, 12 Wks Sofosbuvir/Ledipasvir (N=20) | B: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9669 (N=20) | C: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9451 (N=20) | D Retx: HCV GT-1, Re-Treatment, 12 Wks Sofosbuvir, Ledipasvir (N=34) | D: HCV GT-1, Tx-relapsed, 12 Wks Sofosbuvir/Ledipasvir (N=14) | E: HCV GT-4, tx Naive/Expd, 12 Wks Sofosbuvir/Ledipasvir (N=21) | F: HCV GT-1, tx Naive/Expd 6 Wks Sofosbuvir/Ledipasvir/GS-9451 (N=50) | G: HCV GT-1, tx Naive, 4 Wks Sofosbuvir, Ledipasvir, GS-9451 (N=25) | H: HCV GT-1, tx Naive, 4 Wks Sofos/Ledip/GS-9451/GS-9669 (N=25)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: HCV GT-1, tx Naive, 12 Wks Sofosbuvir/Ledipasvir (N=20) | B: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9669 (N=20) | C: HCV GT-1, tx Naive, 6 Wks Sofosbuvir/Ledipasvir/GS-9451 (N=20) | D Retx: HCV GT-1, Re-Treatment, 12 Wks Sofosbuvir, Ledipasvir (N=34) | D: HCV GT-1, Tx-relapsed, 12 Wks Sofosbuvir/Ledipasvir (N=14) | E: HCV GT-4, tx Naive/Expd, 12 Wks Sofosbuvir/Ledipasvir (N=21) | F: HCV GT-1, tx Naive/Expd 6 Wks Sofosbuvir/Ledipasvir/GS-9451 (N=50) | G: HCV GT-1, tx Naive, 4 Wks Sofosbuvir, Ledipasvir, GS-9451 (N=25) | H: HCV GT-1, tx Naive, 4 Wks Sofos/Ledip/GS-9451/GS-9669 (N=25)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 1 | 0 | 3 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 6 | 3 | 0 | 1 | 3 | 4 | 1 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 0 | 2 | 5 | 0 | 8
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 4 | 2 | 0 | 3 | 6 | 4 | 4
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Urethritis trichomonal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | 2 | 0 | 0 | 8 | 1 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 5 | 0 | 1 | 11 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 2 | 3 | 0 | 0 | 9 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Blood bicarbonate abnormal (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 4 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 5 | 0 | 1 | 2 | 2 | 0 | 3
Blood cholesterol increased (Investigations) | 4 | 3 | 3 | 17 | 3 | 5 | 4 | 7 | 5
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 4 | 6 | 2 | 3 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 3 | 0 | 0 | 1 | 6 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 2 | 4 | 0 | 1
Low density lipoprotein increased (Investigations) | 2 | 2 | 0 | 10 | 3 | 5 | 3 | 5 | 4
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 1 | 1 | 3 | 1 | 2 | 3 | 2 | 3
Platelet count decreased (Investigations) | 3 | 1 | 2 | 1 | 0 | 2 | 5 | 0 | 0
Tuberculin test positive (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 3 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 9 | 9 | 12 | 6 | 8 | 20 | 6 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4 | 0 | 0 | 2 | 2 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 8 | 8 | 0 | 2 | 2 | 3 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 4 | 1 | 2 | 4 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 4 | 0 | 1 | 2 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 6 | 4 | 8 | 2 | 6 | 5 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 6
Headache (Nervous system disorders) | 5 | 5 | 0 | 1 | 2 | 2 | 4 | 1 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spermatocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ex-tobacco user (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Supplementation therapy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Transfusion (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No